CLINICAL TRIAL: NCT07181889
Title: Oxidative Stress and Antioxidant Enzyme Activities in Elite Female Turkish Cross-Country Skiers
Status: Completed | Type: Observational
Sponsor: Duvenciler Anadolu Lİsesi (Other)
Responsible Party: Principal Investigator, Omer Faruk Bilici, Principal Investigator, Duvenciler Anadolu Lİsesi
Other Study IDs: 27754
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Oxidative Stress; Redox Imbalance; Exercise-Induced Physiological Stress
Keywords: Catalase; Glutathione; Malondialdehyde; Oxidative Stress Biomarkers; Endurance Training; Female Athletes; Sports Science

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples obtained from fasting venous blood draws will be retained at -80 °C for future biochemical analysis of oxidative stress and antioxidant biomarkers. No genetic or DNA-based testing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elite Cross-Country Skiers: Female athletes aged 15-20 years who are members of the Turkish junior or senior national cross-country skiing teams. Participants are engaged in regular endurance training and competition. No experimental intervention is applied; participants undergo anthropometric measurements and venous blood sampling for oxidative stress and antioxidant biomarker analysis.
- Sedentary Control Group: Healthy women aged 15-20 years, matched for age and BMI to the athlete group. Participants have no history of regular exercise training for at least 6 months prior to enrollment. No experimental intervention is applied; participants undergo the same anthropometric and blood sampling procedures as the athlete group.

SUMMARY:
This study is designed to investigate oxidative stress and antioxidant defense biomarkers in elite female cross-country skiers compared with sedentary women. Oxidative stress plays a central role in exercise adaptation, and the balance between reactive oxygen species production and antioxidant capacity can influence performance and recovery. Despite growing interest in redox biology, evidence from elite female endurance athletes is limited.

This cross-sectional observational study enrolled 17 elite female cross-country skiers, who were members of the Turkish national junior and senior teams, and 17 age- and BMI-matched sedentary women. All participants reported to the laboratory between 07:00 and 09:00 a.m. after an overnight fast. Anthropometric characteristics, including height, weight, and BMI, were measured under standardized conditions.

Venous blood samples were collected from the antecubital vein using aseptic technique. Serum was separated, stored at -80 °C, and analyzed for key redox biomarkers. Catalase (CAT) activity was measured spectrophotometrically using the method of Aebi, reduced glutathione (GSH) concentration was determined using Ellman's reagent, and malondialdehyde (MDA), a marker of lipid peroxidation, was assessed using the thiobarbituric acid reactive substances (TBARS) assay. All analyses were performed in triplicate in a certified clinical biochemistry laboratory.

The primary objective of this study is to characterize and compare systemic antioxidant capacity and oxidative stress levels between trained athletes and sedentary controls. The data generated will provide insight into how chronic endurance training in cold outdoor environments affects enzymatic and non-enzymatic antioxidant systems in young women.

DETAILED DESCRIPTION:
This study was designed as a cross-sectional observational investigation to examine systemic oxidative stress and antioxidant defenses in elite female cross-country skiers compared with sedentary women of similar age and body mass index. The study followed the STROBE guidelines for reporting observational research and complied with the principles of the Declaration of Helsinki. Ethical approval was granted by the Muş Alparslan University Scientific Research and Publication Ethics Committee (Approval No: 27754; Date: 27 October 2021).

Participants

A total of 34 women participated in the study, including 17 elite female cross-country skiers who were current members of the Turkish national junior and senior teams (2021-2025 competitive seasons) and 17 sedentary women matched for age and BMI. Inclusion criteria were: (a) female sex; (b) age between 15-20 years; (c) absence of chronic metabolic, cardiovascular, or inflammatory diseases; (d) no regular medication use; (e) no vitamin or antioxidant supplementation within the preceding three months; and (f) non-smoker and non-alcohol consumer. Exclusion criteria included acute infection, recent musculoskeletal injury, or failure to comply with pre-test requirements (e.g., overnight fasting, rest). Written informed consent was obtained from all participants; for those under 18 years of age, parental or guardian consent was also collected.

Anthropometric and Pre-Analytical Procedures

All participants attended the laboratory between 07:00 and 09:00 a.m. following a 10-12-hour overnight fast to minimize the effect of circadian variation and dietary intake on oxidative stress markers. Upon arrival, participants were asked to remain seated in a quiet, temperature-controlled room (22-24 °C) for at least 30 minutes to achieve resting physiological conditions. Anthropometric measurements were taken barefoot and in light clothing using standardized procedures: standing height was measured to the nearest 0.1 cm using a stadiometer, and body weight was measured to the nearest 0.1 kg with a calibrated digital scale. Body mass index (BMI) was calculated as weight (kg) divided by height squared (m²).

Blood Sampling and Processing

Venous blood samples (approximately 3 mL) were collected from the antecubital vein using sterile vacutainer tubes. Samples were allowed to clot for 20-30 minutes at room temperature and subsequently centrifuged at 5000 rpm for 10 minutes to separate serum. Serum aliquots were transferred into labeled polypropylene tubes and stored at -80 °C until biochemical analysis. Previous studies have confirmed the stability of oxidative stress biomarkers, including reactive oxygen metabolites and antioxidant potential, in serum stored under these conditions for up to five years.

Biochemical Analyses

All analyses were performed in the Central Biochemistry Laboratory of Van Yüzüncü Yıl University Faculty of Medicine by the same experienced laboratory technician to minimize inter-operator variability.

Catalase (CAT) activity was determined according to the spectrophotometric method of Aebi, which measures the rate of hydrogen peroxide decomposition at 240 nm over a two-minute interval at 25 °C. Results were expressed as units per milliliter (U/mL).

Reduced Glutathione (GSH) concentration was quantified using the colorimetric method of Beutler et al., employing Ellman's reagent (5,5'-dithiobis-(2-nitrobenzoic acid), DTNB) to produce a yellow-colored compound measurable at 412 nm.

Malondialdehyde (MDA) concentration, a marker of lipid peroxidation, was measured by the thiobarbituric acid reactive substances (TBARS) assay, based on the formation of a pink MDA-TBA complex read at 532 nm.

Each sample was analyzed in triplicate, and mean values were used for subsequent statistical processing to increase measurement reliability.

Data Management and Planned Analyses

Data were entered into a secure electronic database and cross-checked for accuracy by two independent researchers. Descriptive statistics (mean ± standard deviation, minimum-maximum) were calculated for all continuous variables. The normality of data distributions was assessed using the Shapiro-Wilk test. For variables not meeting the assumption of normality, non-parametric tests (Mann-Whitney U test) were pre-specified to compare group differences. Effect sizes were to be calculated using Cohen's d with 95% confidence intervals to quantify the magnitude of between-group differences. Correlations between CAT, GSH, and MDA were planned using Spearman rank-order correlation coefficients. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 15-20 years
* Members of the Turkish junior or senior national cross-country skiing team (for athlete group)
* Sedentary lifestyle, no regular exercise training within the past 6 months (for control group)
* Body mass index within normal range (18.5-24.9 kg/m²)
* No use of antioxidant or vitamin supplementation within the past 3 months
* Non-smoker and no alcohol consumption
* Voluntary participation with signed informed consent (and parental consent if under 18 years)

Exclusion Criteria:

* Presence of chronic metabolic, cardiovascular, or inflammatory diseases
* Current medication use affecting oxidative stress or metabolism
* Acute infection or illness within 2 weeks prior to data collection
* Recent musculoskeletal injury or inability to comply with testing procedures
* Failure to complete overnight fasting or rest requirements before blood sampling

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study included 34 healthy female participants: 17 elite cross-country skiers and 17 sedentary controls matched for age and BMI. All participants were aged 15-20 years and met strict inclusion and exclusion criteria to ensure a homogeneous sample.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Serum Catalase (CAT) Activity | Baseline (single fasting blood draw)
  Catalase activity in serum measured spectrophotometrically at 240 nm following Aebi's method; expressed as units per milliliter (U/mL).
Serum Reduced Glutathione (GSH) Concentration | Baseline (single fasting blood draw)
  Total glutathione concentration measured colorimetrically using Ellman's reagent (DTNB); expressed as µmol/L.
Serum Malondialdehyde (MDA) Concentration | Baseline (single fasting blood draw)
  Marker of lipid peroxidation measured via thiobarbituric acid reactive substances (TBARS) method; expressed as nmol/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Faculty of Sports Sciences, Muş, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive personal health information and the sample size is small, which may compromise participant confidentiality.